CLINICAL TRIAL: NCT01604304
Title: Flexible urétéroscopy Versus Extracorporeal Shockwave Lithotripsy in 5 to 20 mm Renal Calculi, Efficacity Prospective Randomized Trial
Brief Title: Flexible urétéroscopy Versus Extracorporeal Shockwave Lithotripsy in Renal Calculi
Acronym: CALIX-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011.692
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2014-08

CONDITIONS: Extracorporeal Shockwave Lithotripsy, Flexible Ureteroscopy
Keywords: stone; calculi; kidney; renal treatment; flexible ureteroscopy; extracoporeal shockwave lithotripsy; retrograde intra renal surgery
MeSH Terms: conditions — Calculi | interventions — Lithotripsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extracorporeal shockwave lithotripsy (Active Comparator): stone treatment using electroconductive technology
  Interventions: Procedure: extracorporeal shockwave lithotripsy
- Flexible ureteroscopy (Active Comparator): intra renal retrograde surgery with or without laser and stone extraction
  Interventions: Procedure: flexible ureteroscopy

INTERVENTIONS:
Procedure: flexible ureteroscopy — Flexible ureteroscopy will be use for 120 min max to treat renal stone. Laser, access sheath, baskets can be use to perform the technique.
  Arms: Flexible ureteroscopy
Procedure: extracorporeal shockwave lithotripsy — The lithotriptor is use with 1,1 Hz frequency and stop when patient get 1000 joules of energy or if there is a problem with tolerance of this treatment or if stone is broken
  Arms: Extracorporeal shockwave lithotripsy

SUMMARY:
Flexible ureteroscopy is a recent procedure to treat renal stone. Extracorporeal shockwave lithotripsy was the gold standard treatment for calculi between 5 and 20 mm. In literature, the two procedures are available to treat these stones with a good stone free rate. There is no prospective randomized study comparing these two treatments. Our study will define with a good level of evidence which technique is the best with regard to the stone free rate, secondary procedure rate and adverse effect.

ELIGIBILITY:
Inclusion Criteria:

* Patient with 5 to 20 mm renal stone
* Age ≥ 18 years old
* Patient agreement signed
* BMI < 35
* Contraception

Exclusion Criteria:

* Pregnancy
* Severe musculoskeletal deformities
* Renal artery or aorta aneurysm
* Pacemaker
* Anesthesia contra indication
* Psychiatric trouble or law protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Stone free rate | Three months
  Rate of stone free patient or patient with residual fragment ≤ 3 mm, 3 months after the treatment evaluated, will be compare. This outcome is measured with a tomodensitometry and compares with pre treatment exams.

SECONDARY OUTCOMES:
Stone free rate in weight's sub group | 3 months
  Each arm wil be divise in 3 sub group based on body mass index (20 to 25, 25 to 30, 30 to 35). We'll compare rate of efficacity in each sub group
Stone free rate in sub group depending on stone diameters | 3 months
  Each arm wil be divise in 3 sub group based on calculi diameter (5 to 10mm, 10 to 15 and 15 to 20). We'll compare rate of efficacity in each sub group
Secondary procedure rate | 3 months
  In each arm will be evaluate rate of secondary procedure needed to have the best stone free rate
Serious and non serious adverse events | 3 months
  In each arm will be evaluate rate of adverse event, type, severity.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Martin, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service d'urologie, Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Result] Ravier E, Abid N, Ruffion A, Fassi-Fehri H, Buron C, Ganne C, Mallet A, Martin X. [Effectiveness of flexible ureteroscopy versus extracorporeal shock wave lithotripsy for kidney stones treatment]. Prog Urol. 2015 Apr;25(5):233-9. doi: 10.1016/j.purol.2015.01.005. Epub 2015 Jan 29. French. PMID 25640027